CLINICAL TRIAL: NCT03413657
Title: Predicting Fluid Responsiveness Using Transiently Increased Intrathoracic Pressure in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 1086731
Record Dates: First submitted 2018-01-11; First posted 2018-01-29 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Fluid Reponsiveness

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either undergo the PEEP challenge or tidal volume challenge first. After the initial challenge, subjects will cross over to whichever challenge has not yet been performed.
  Subjects will be separated into the following categories: "fluid responders" and "non-responders" and analyzed in those categories.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid responders (Other): Patient's identified to have a significant increase in their cardiac output following a fluid bolus.
  Interventions: Procedure: Increase in intrathoracic pressure
- Fluid non-responders (Other): Patient's identified to NOT have a significant increase in their cardiac output following a fluid bolus.
  Interventions: Procedure: Increase in intrathoracic pressure

INTERVENTIONS:
Procedure: Increase in intrathoracic pressure — Will transiently increase intrathoracic pressure for 60 seconds and monitor for changes in hemodynamics during this time.
  Other Names: PEEP Challenge; Tidal Volume Challenge

SUMMARY:
The goal of this study is to identify in patients requiring active fluid resuscitation and mechanical ventilation for circulatory shock, can a controlled increase in intrathoracic pressure (either by positive-end expiratory pressure (PEEP) or tidal volume (TV)) predict responsiveness to additional fluid resuscitation.

We hypothesize that a temporary, physiologically-safe increase in positive-end expiratory pressure (PEEP) and/or a temporary increase in tidal volume (from 6 cc/kg predicted body weight (PBW) to 8 cc/kg PBW) in patients requiring invasive mechanical ventilation will predict fluid responsiveness based upon an assessment of the change in pulse pressure and stroke volume variation.

DETAILED DESCRIPTION:
Once an eligible subject is identified and written or telephone consent is obtained from the patient or surrogate as appropriate, we will record demographic data and clinical information including age, sex, height, actual body weight, predicted body weight (PBW), APACHE II on admission, primary diagnosis, reason for ICU admission, and dose of vasopressors.

Patients will be intubated and on assist-control volume ventilation receiving low tidal volumes. Sedation will be titrated per current MICU protocol to minimize patient discomfort and minimizing ventilator dyssynchrony. In keeping with standard practice, the dose of vasoactive medications will be kept constant during the intervention period. The standard practice is to titrate vasopressor therapy every five minutes, so keeping vasoactive medications constant for sixty seconds is in keeping with the standard of care. All subjects will be in an ICU setting and monitored per standard of care (vital signs, telemetry, ventilator data) by a respiratory therapist, pulmonary and critical care fellow or faculty member, and critical care nurse at the bedside throughout the entire intervention.

A point of care (POC) echocardiogram will be performed by the investigator performing the intervention in order to measure the stroke volume index (surrogate for cardiac output).

Subjects will be randomized to either undergo the PEEP challenge or tidal volume challenge first. After the initial challenge, subjects will cross over to whichever challenge has not yet been performed.

The simple changes to the ventilator we are proposing to use as challenges in this study are done frequently and routinely in the ICU with or without the supervision of a physician, but we will have a physician present throughout the entire proposed intervention. For the subjects undergoing PEEP challenge first, we will do the following:

1. POC echocardiogram performed to measure SVI
2. The tidal volume will be set to 6 mL/kg PBW and the patients will be monitored for 5 minutes for any variability in vital parameters. The subject's ventilatory parameters, vitals, hemodynamics, and oxygenation will be recorded on initial ventilator settings.
3. PEEP challenge - PEEP will be increased by 50% for 60 seconds. The subject's ventilatory parameters, vitals, hemodynamics, and oxygenation will be recorded after 60 seconds.
4. PEEP returned to initial settings.
5. 2 minute washout period to prepare for tidal volume challenge.
6. Tidal volume challenge - tidal volume raised to 8 cc/kg PBW for 60 seconds. The subject's ventilatory parameters, vitals, hemodynamics, and oxygenation will be recorded will be recorded after 60 seconds.
7. Subjects ventilator settings returned to initial settings x 2 minutes.
8. 500 cc crystalloid fluid bolus of the ICU team's choosing is then administered to the patient. The subject's ventilatory parameters, vitals, hemodynamics, and oxygenation will be measured.
9. POC echocardiogram performed to measure SVI and determine if the subject is a fluid responder or non-responder.

The procedure for those randomized into the tidal volume challenge first will be similar, but the tidal volume challenge (e, above), rather than the PEEP challenge (b, above), will be performed first.

In the management of a critically ill patient in circulatory shock, physicians encounter the question of whether to administer fluid to the patient or not several times during the course of the patient's stay in the ICU. To ensure that our study is generalizable and applicable, we will perform the above protocol up to three times per subject. This is similar to previous studies using changes in intrathoracic pressure to predict fluid responsiveness. Additionally, we will have a larger number of interventions in order to better show a clear difference statistically.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated
* Identified by treatment team as requiring intravenous fluid bolus
* Acute circulatory failure during admission (systolic blood pressure (SBP) ≤90 mmHg or mean arterial pressure (MAP) ≤70 mmHg or requiring vasopressors to maintain SBP >90 mmHg or MAP >70 mmHg, along with one or more of the following:
* urinary flow ≤0.5 mL/kg/min for ≥2 hours,
* heart rate ≥100 beats per minute
* presence of skin mottling
* blood lactate concentration ≥4 mmol/L

Exclusion Criteria:

* Contraindication to fluid bolus
* Assynchrony Index > 10%
* Clinically significant cardiac arrhythmia
* Severe valvular heart disease
* Chest tubes with air leak
* Abdominal compartment syndrome
* Pregnancy
* Concurrent nebulized medication or inhaled nitric oxide
* Transthoracic echogenicity unsuitable for measuring velocity-time integral of aortic blood flow (SVI)
* Prisoner
* Clinical brain death
* PEEP > 15 cmH2O

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Pulse Pressure Variation | Following 60 seconds of intrathoracic pressure challenge
  Temporary increase in intrathoracic pressure (PEEP or TV) will predict fluid responsiveness using an absolute increase in pulse pressure variation by 3% or more.

SECONDARY OUTCOMES:
Heart Rate | Following 60 seconds of intrathoracic pressure challenge
  Temporary increase in intrathoracic pressure (PEEP or TV) will predict fluid responsiveness using an absolute decrease in heart rate by 15 beats per minute or more.
Mean Arterial Pressure | Following 60 seconds of intrathoracic pressure challenge
  Temporary increase in intrathoracic pressure (PEEP or TV) will predict fluid responsiveness using an absolute decrease in MAP by 15 mmHg or more.
Mortality | 7 days
  Differences in 7 day mortality between fluid responders and non-responders
Stroke Volume Variation | Following 60 seconds of intrathoracic pressure challenge
  Temporary increase in intrathoracic pressure (PEEP or TV) will predict fluid responsiveness using an absolute increase in SVV of 4% or more.
End-tidal carbon dioxide | Following 60 seconds of intrathoracic pressure challenge
  Temporary increase in intrathoracic pressure (PEEP or TV) will predict fluid responsiveness using an increase in EtCO2 by 4% or more.

CONTACTS AND LOCATIONS:
Overall Officials: John Adams, MD, Principal Investigator — Attending Physician
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided